CLINICAL TRIAL: NCT07104123
Title: Substance Use in Pregnant People - Optimizing Retention in Treatment by Maximizing Opportunities for Management
Brief Title: Substance Use in Pregnant People - Optimizing Retention in Treatment
Acronym: SUPPORT-MOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R61DA062321 (NIH); R61DA062321 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Substance Use Disorder (SUD); Pregnancy; Postpartum; Contingency Management
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social drivers of health screening (Experimental)
  Interventions: Other: Social drivers of health screening
- Contingency Management (Experimental)
  Interventions: Behavioral: Patients will undergo a program of contingency management

INTERVENTIONS:
Other: Social drivers of health screening — Patients will undergo a structured and protocoled screening for social drivers of health and be linked to support services
  Arms: Social drivers of health screening
Behavioral: Patients will undergo a program of contingency management — Patients will enter into a 12 week program of contingency management
  Arms: Contingency Management

SUMMARY:
Substance use during pregnancy is a leading cause of maternal morbidity and mortality in the United States, with 55-80% of postpartum patients disengaging from substance use disorder (SUD) treatment within one year of delivery. Structural and social determinants of health, including housing instability, transportation barriers, and limited childcare access, further exacerbate disparities in treatment retention.

This pilot study, conducted in two specialized prenatal care clinics, evaluates the feasibility and acceptability of two integrated strategies to promote sustained engagement in recovery-oriented services during the perinatal and postpartum periods. Aim 1 implements a standardized social needs screening and referral protocol to connect patients with community-based supports. Aim 2 pilots a contingency management intervention to incentivize recovery-supportive behaviors.

Findings will inform the design of a larger multi-site randomized controlled trial to evaluate the impact of these interventions on treatment retention, overdose prevention, and maternal-infant health outcomes.

DETAILED DESCRIPTION:
Substance use during pregnancy remains a significant public health concern and is among the leading causes of maternal morbidity and mortality in the United States. Despite the availability of evidence-based interventions-including pharmacotherapy and behavioral counseling-treatment discontinuation in the postpartum period remains prevalent. Data from prior studies indicate that between 55% and 80% of postpartum patients disengage from substance use disorder (SUD) treatment within the first year following delivery. Disparities in treatment retention are further exacerbated by structural and social determinants of health, such as housing instability, transportation barriers, and limited access to childcare.

This pilot study is conducted in two specialized prenatal care clinics for individuals with SUD. The primary objective is to evaluate the feasibility and acceptability of two integrated, patient-centered strategies designed to promote sustained engagement in recovery-oriented services during the perinatal and postpartum periods.

Aim 1: Implementation of a Standardized Social Needs Screening and Referral Protocol This aim assesses the feasibility of deploying a structured, clinic-based protocol to systematically identify and address unmet social needs among pregnant patients with SUD. The protocol includes referral pathways to community-based services, including but not limited to perinatal home visiting programs, doulas, housing assistance, and transportation resources. Approximately 20 patients receiving care in the CARE clinic are enrolled to evaluate the clarity, usability, and clinical integration of the screening and referral process.

Aim 2: Pilot Testing of a Contingency Management Intervention This aim pilots a contingency management framework to incentivize engagement in recovery-supportive behaviors, such as attending scheduled appointments, adhering to treatment plans, and participating in supportive health activities. Contingency management demonstrates efficacy in other populations but has not been sufficiently adapted for use in perinatal SUD treatment settings. Approximately 20 patients are enrolled in this arm to assess the feasibility, fidelity, and preliminary acceptability of the intervention.

Both components of the study are designed to enhance long-term maternal recovery outcomes by delivering tailored, real-world supports that extend beyond delivery into the vulnerable postpartum period. Insights gained from this pilot study inform the development of a larger, multi-site randomized controlled trial to rigorously evaluate the impact of the interventions on treatment retention, overdose risk reduction, and maternal-infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Confirmed viable intrauterine pregnancy at any gestational age, or within three years postpartum

SUD as defined in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders or clinician documentation

Exclusion Criteria:

Decline follow-up care at study site

Require immediate hospitalization for unstable medical or psychiatric conditions making them clinically unsuitable to participate in a research study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Social Drivers: Enrollment | Enrollment Visit
  Percentage of eligible patients enrolled in the study
Social Drivers: Screening | Through study completion, up to six months postpartum
  Percentage of visits for enrolled patients with social drivers of health screening
Social Drivers: Documentation of Z-codes | Through study completion, up to six months postpartum
  Percentage of social driver screenings with z-codes documented
Contingency Management: Intervention Fidelity (Number of Visits) | Weekly from enrollment up to 12 weeks
  Number of CM sessions with fidelity to intervention, defined as meeting all six criteria on weekly CM visit checklist
Contingency Management: Intervention Fidelity (Percentage of Visits) | Weekly from enrollment up to 12 weeks
  Percentage of CM sessions with fidelity to intervention, defined as meeting all six criteria on weekly CM visit checklist
Contingency Management: Acceptability of Intervention Measure (AIM) | After 3 CM sessions (up to 3 weeks), end of intervention (up to 12 weeks)
  Weiner et al, Implement Sci, 2017
Contingency Management: Intervention Appropriateness Measure (IAM) | After 3 CM sessions (up to 3 weeks), end of intervention (up to 12 weeks)
  Weiner et al, Implement Sci, 2017
Contingency Management: Feasibility of Intervention Measure (FIM) | After 3 CM sessions (up to 3 weeks), end of intervention (up to 12 weeks)
  Weiner et al, Implement Sci, 2017

SECONDARY OUTCOMES:
Social Drivers: Frequency of Z-Codes | End of intervention (up to 12 weeks postpartum)
  Frequency of of z-codes documented for each patient
Social Drivers: Percentage of Patients with Referrals | End of intervention (up to 12 weeks postpartum)
  Percentage of patients with referrals to support services

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie C Kelly, MD, MS, Principal Investigator — Washington University School of Medicine; Ana Baumann Walker, PhD, MA, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
NICHD Data and Specimen Hub (DASH)
Supporting Information: Study Protocol
Time Frame: Start Date: 9/1/2025 End Date: 8/31/2028
Access Criteria: Authorized users will access the data through the NICHD Data and Specimen Hub (DASH) repository and the NIH HEAL Initiative Data Platform
URL: https://healdata.org/portal/discovery/HDP01415/